CLINICAL TRIAL: NCT00171496
Title: A Six-month Open Label, Multicenter, Randomized Study to Evaluate the Incidence of New Onset Diabetes Mellitus and Glucose Metabolism in Patients Receiving Cyclosporine Microemulsion With C-2 Monitoring Versus Tacrolimus After de Novo Kidney Transplantation
Brief Title: Evaluation of Cyclosporine Microemulsion and Tacrolimus on the Rate of New Onset Diabetes Mellitus in Kidney Transplantation Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COLO400A2419
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Transplant
Keywords: Kidney transplant, adults, NODM, immunosuppressants
MeSH Terms: interventions — Tacrolimus

ARMS (2):
- Cyclosporine microemulsion (Experimental)
  Interventions: Drug: Cyclosporine microemulsion
- Tacrolimus (Active Comparator)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Cyclosporine microemulsion
  Arms: Cyclosporine microemulsion
Drug: Tacrolimus
  Arms: Tacrolimus

SUMMARY:
The purpose of this study is to evaluate the impact of tacrolimus and cyclosporine microemulsion on glucose metabolism in kidney transplant recipients and the efficacy and safety in preventing organ rejection

ELIGIBILITY:
Inclusion Criteria:

- First or second transplant, cadaveric or living donor

Exclusion Criteria:

* Multi-organ or dual kidney transplants
* Panel reactive antibodies >50%

Other protocol-defined inclusion/exclusion criteria applied

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 693 (Actual)
Dates: Start 2003-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Incidence of NODM or impaired fasting glucose (IFG) in de novo kidney transplant patients receiving cyclosporine microemulsion versus in patients receiving tacrolimus within the first 6 months post-transplantation.
Incidence of biopsy-proven acute rejection (BPAR) or graft loss or death within the first 6 months post-transplantation.

SECONDARY OUTCOMES:
incidence of NODM or IFG within the first 3 mths post-transplantation in pts treated with cyclosporine microemulsion or tacrolimus
percentage of pts with preexisting diabetes at transplantation who have a glycosylated hemoglobin level >7% at Mths 3 &6 post-transplantation
Change over time of mean HbA1c at mths 3 &6 post-transplantation in pts w/ preexisting diabetes at transplantation
percentage of pts who switched from oral hypoglycemic agents to insulin within 3 &6 mths post-transplantation
incidence of impaired glucose tolerance (IGT) as assessed by an oral glucose tolerance test (OGTT) | 6 months
Blood pressure at Months 3& 6 post-transplantation
incidence of BPAR or graft loss or death within the first 3 months post-transplantation, as well as the incidence of each individual event within 3 and 6 months post-transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis

REFERENCES:
- [Result] Ekmekcioglu O, Turkan S, Yildiz S, Gunes ZE. Comparison of tacrolimus with a cyclosporine microemulsion for immunosuppressive therapy in kidney transplantation. Turk J Urol. 2013 Mar;39(1):16-21. doi: 10.5152/tud.2013.004. PMID 26328072